CLINICAL TRIAL: NCT05715112
Title: Graded Motor Imagery and Fall Risk in Older Adults: An Exploratory Study
Brief Title: Graded Motor Imagery and Fall Risk in Older Adults
Acronym: GMI
Status: Completed | Type: Observational
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Professor Emeritus / Principal Investigator, St. Ambrose University
Other Study IDs: StAmbroseU GMI fall risk
Record Dates: First submitted 2023-01-13; First posted 2023-02-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Balance; Fall Risk
Keywords: Graded Motor Imagery; Balance; Fall Risk; Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: A convenience sample of older adults (65 and older).
  Interventions: Procedure: Graded Motor Imagery

INTERVENTIONS:
Procedure: Graded Motor Imagery — GMI consisting of education, sensory integration of the foot using contact, flooring samples, immersion, and two point discrimination.
  Other Names: GMI

SUMMARY:
To determine if there is any carry over effect of sensation training for the feet, officially called Graded Motor Imagery (GMI), will impact balance and fall risk factors in older individuals. This will be looked at to see if there is a difference in balance and sensation before and right after the training.

DETAILED DESCRIPTION:
In order to increase acuity of body maps, various tactile and movement-based strategies have been recommended and supported for research focusing on sensory discrimination. Current evidence, specific to painful conditions related to altered cortical mapping, have shown growing evidence in reducing pain and disability. In regards to it's ability to alter foot pain in older adults and decreasing fall risk, prior conference case study and case series presentations have suggested potential clinical benefit, but it has not been formally studied. The aim of this study is to determine if a sensory discrimination training for feet in older adults can alleviate pain, improve sensory discrimination, and also decrease fall risk. Specifically, does a 20 minute training session improve pain, balance (Brief-BEST test), and sensory discrimination in individuals over 65 years of age. Secondary analysis may exam characteristics that best identify those who benefit from this training.

ELIGIBILITY:
Inclusion Criteria:

* Be able to read and understand English
* Be over the age of 65
* Be independent with ambulation (with or without an assistive device)
* Not have any skin condition or injury to the plantar or dorsal part of the foot
* Have the visual ability to view images on a tablet to partake in a test

Exclusion Criteria:

* No existing skin conditions on the bottom of the foot that would impair sensation
* No current injury to the plantar or dorsal side of the foot
* No prior surgery or major injury to the plantar or dorsal side of the foot
* Lacking sensation in the foot
* Unable to read and understand English
* Lacking ability to view images on a tablet to partake in a test
* Unable to ambulate (with or without an assistive device)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A convenience sample of older adults (65 and older) will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Lower extremity pain rating | self-reported, change from before to immediately after treatment
  Change (from before treatment to immediately after treatment) in pain for the lower extremity using the numeric pain rating scale (NPRS - 0 to 10 where 0 = no pain and 10 + maximum pain)
Laterality Speed | tested for 60 seconds before and immediately after treatment
  Change (from before treatment to immediately after treatment) in speed of foot recognition using Recognize (TM) (speed in seconds to recognize each of 40 images as right or left foot)
Laterality Accuracy | tested for 60 seconds before and immediately after treatment
  Change (from before treatment to immediately after treatment) in accuracy of foot recognition using Recognize (TM) (percent accurately correctly identified as right or left foot of those 40 images)
Balance / fall risk | Assessed before and immediately after treatment
  Change (from before treatment to immediately after treatment) in Brief-BESTest (6 task subsets to assess static and dynamic balance) (0 - 15 scale where 0 - lowest score / unstable and 15 = highest / no balance issues)
Nerve Sensitivity Dorsum of dominant hand | Assessed before and immediately after treatment
  Change (from before treatment to immediately after treatment) in Pain Pressure Threshold (PPT) on dorsum of web space of dominant hand (in pounds)
Nerve Sensitivity Dorsum of Right Foot | Assessed before and immediately after treatment
  Change (from before treatment to immediately after treatment) in Pain Pressure Threshold (PPT) on dorsum of right foot (in pounds)
Nerve Sensitivity Dorsum of Left Foot | Assessed before and immediately after treatment
  Change (from before treatment to immediately after treatment) in Pain Pressure Threshold (PPT) on dorsum of left foot (in pounds)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, PT, PhD, Principal Investigator — St. Ambrose University
Locations (1):
- St. Ambrose University, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No